CLINICAL TRIAL: NCT06231225
Title: Study on the Effect of Incentive Spirometer-based Respiratory Training on the Long COVID-19 Symptoms in Chronic Disease Patients After Recovery From COVID-19
Brief Title: Study on the Effect of Incentive Spirometer-based Respiratory Training on the Long COVID-19
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yu-Shan Hsieh, Assistant professor, National Taipei University of Nursing and Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B202305165
Record Dates: First submitted 2024-01-26; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: COVID-19 Pandemic; Diabetes; Hypertension; Cardiac Disease; Long COVID
Keywords: COVID-19; Post-Acute COVID-19 Syndrome; Long COVID-19; respiratory training; Hypertensive diseases; Cardiac diseases; Diabetes; Dyspnea; Incentive Spirometer
MeSH Terms: conditions — COVID-19; Diabetes Mellitus; Hypertension; Heart Diseases; Post-Acute COVID-19 Syndrome; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): not assign respiratory training
- treatment group (Experimental): assign respiratory training
  Interventions: Behavioral: Incentive Spirometer respiratory training

INTERVENTIONS:
Behavioral: Incentive Spirometer respiratory training — The incentive spirometer is a handheld mechanical breathing device that uses a one-way valve to prevent exhalation. It consists of a corrugated tube and a nozzle connected to three consecutive plastic chambers, each containing a ball. The external chambers are marked with the minimum flow required to raise the ball internally. The ball rises when the patient performs slow, deep breathing through the nozzle. If the patient breathes too quickly, the balls in the chambers rise to the top, and if breathing is too slow, the balls fall to the bottom. The number of increasing balls measures the volume of inhaled air. When all three balls reach the top of the chambers, the patient's flow rate can reach 1200 ml/s. After the patient has maximized their inhalation, they are asked to hold the balls in the same position for more than 3 sec.
  Arms: treatment group

SUMMARY:
The COVID-19 pandemic has emerged as the most significant public health crisis of the 21st century. As of the end of January 2023, global confirmed cases have exceeded 670 million, with a domestic cumulative total of 10.24 million cases, including occurrences of reinfection. Beyond acute symptoms following infection, patients and society face the challenge of long-term complications associated with COVID-19. Termed 'Post COVID-19 condition' or 'Long COVID' by the World Health Organization (WHO), this encompasses symptoms appearing within three months of the initial infection. Symptoms of Long COVID reveal chronic damage inflicted by the virus on multiple organ systems, including fatigue, cognitive impairment, chest tightness, palpitations, difficulty breathing, and depression.

Despite continuous efforts by healthcare professionals to find suitable treatments, no medication has been confirmed to effectively prevent or reduce post-COVID-19 sequelae. These health issues impose significant burdens and disturbances on patients' quality of life, economies, and societies.

DETAILED DESCRIPTION:
According to the Ministry of Health and Welfare's report on the top 10 causes of death in the 111th year, aside from the marked increase in COVID-19 cases, there have been significant increases in hypertensive diseases, Cardiac diseases, and diabetes .Therefore, addressing the post-COVID-19 sequelae among chronic disease patients is an essential global health issue in the post-pandemic era.

Current research indicates that respiratory training is safe and effective in improving the exercise capacity, lung function, and alleviating respiratory difficulties in COVID-19 recovered patients. The impact of respiratory training on patients' respiratory and physical function remains uncertain, especially considering that many present-day infections are among non-hospitalized individuals with mild symptoms. Thus, exploring simple and effective respiratory training methods to reduce COVID-19's long-term impact on patients warrants continuous investigation.

Therefore, this study will employ Incentive spirometer-based respiratory training to assist COVID-19 patients who has diabetes, hypertensive disease, or cardiac disease in respiratory training. Data collection before and after the intervention will involve oxygen demand, blood parameters, the post-COVID-19 Functional Status scale (PCFS scale), and lung function indices, to investigate and evaluate the effectiveness of intervention respiratory training in improving Long COVID symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who have contracted and recovered from COVID-19 within the past year must present proof of diagnosis, such as medical certificates or screening results. The ICD-10 diagnosis codes are: U07.1 for confirmed COVID-19 viral infection, and U09.0 for post-COVID-19 condition, unspecified. Recovery is defined as testing negative in a COVID-19 rapid test.
2. Never diagnosed with hypertensive diseases (ICD-10 codes: I10.x or I11.x), diabetes (ICD-10 codes: E10.x or E11.x), or heart diseases (ICD-10 codes: I25.x, I50.x, I65.x, or I67.x and classified as Class I or II by the New York Heart Association functional classification).
3. Exhibiting long-term respiratory symptoms related to COVID-19, such as post-exertional breathlessness, chest discomfort, cough, difficulty breathing, rapid breathing, etc., and meeting at least one of these criteria for inclusion.
4. Aged between 20 - 90 years.
5. Able to communicate in and understand Mandarin or Taiwanese, either verbally or non-verbally.
6. Willing to participate in the study and agree to be assigned.

Exclusion Criteria:

1. Patients with a functional status classified as level 5 or higher on the Modified Rankin Scale (MRS), indicating severe disability and bedridden status.
2. Patients suffering from dementia, such as Alzheimer's, Parkinson's disease, etc.
3. Patients with acute psychiatric symptoms who are unable to communicate.
4. Individuals with a high risk of litigation.
5. Patients suffering from Chronic Obstructive Pulmonary Disease (COPD) or any other respiratory system diseases.
6. Patients with moderate or severe heart disease, classified as Class III or IV by the New York Heart Association functional classification.

   -

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Post-COVID-19 Functional Status scale | through study completion, an average of 1 year
  for check the effect of respiratory training

SECONDARY OUTCOMES:
Lung function indices | through study completion, an average of 1 year
  for check the effect of respiratory training
Hemoglobin and oxygen levels | through study completion, an average of 1 year
  for check the effect of respiratory training
Six-minute walk test (6MWT) | through study completion, an average of 1 year
  for check the effect of respiratory training
Dyspnoea-12 (D-12) scale | through study completion, an average of 1 year
  for check the effect of respiratory training

IPD SHARING:
Plan to Share IPD: No